CLINICAL TRIAL: NCT05174767
Title: A ProspEctive, Single ARm, Multi-center Clinical InveStigation to EValuatE the Safety and Effectiveness of AMDS in the TREatment of Acute DeBakey Type I Dissection: PERSEVERE
Brief Title: PERSEVERE- a Trial to Evaluate AMDS in Acute DeBakey Type I Dissection
Acronym: PERSEVERE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artivion Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMDS2101.000-C (02/21)
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Acute Aortic Dissection
Keywords: Aortic Diseases; Cardiovascular Diseases; Aortic Dissection; Aortic Remodeling; Malperfusion; Acute; Acute Aortic Dissection
MeSH Terms: conditions — Aortic Diseases; Cardiovascular Diseases; Aortic Dissection

STUDY DESIGN:
Intervention Model Description: Primary Cohort (n=93) and Continued Access (n=40)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Acute DeBakey Type I Dissection (Experimental): In eligible patients, the ascending aorta is transected and removed in a routine standard of care manner utilizing hypothermic circulatory arrest; the operator will leave at least 10 mm (1.0 cm) aortic tissue proximal to the innominate artery. AMDS is pre-loaded onto the delivery system and is delivered into the true lumen through the open distal aorta and implanted according to the instructions for use.
  Interventions: Device: AMDS

INTERVENTIONS:
Device: AMDS — AMDS Implantation

SUMMARY:
Prospective, non-randomized, multicenter clinical investigation to assess the safety and effectiveness of AMDS in the treatment of patients with acute DeBakey type I dissection, with evidence of malperfusion, through open surgical repair.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age or ≤80 years of age (male or female) at time of surgery
* Acute DeBakey type I dissection based on computed tomography angiography (CTA) and diagnosed ≤14 days from of the index event
* Presence of malperfusion (cerebral, visceral, renal, spinal cord, and/or peripheral)

Exclusion Criteria:

* Other medical condition that is associated with limited life expectancy <2 years (e.g., cancer, congestive heart failure)
* Pregnant or breastfeeding.
* Unwilling to comply with the follow-up schedule
* Institutionalized due to administrative or judicial order
* Unwilling to accept blood transfusions for any reason
* Coronary malperfusion
* In circulatory shock (i.e., systolic blood pressure <90 mmHg) at time of screening
* In extreme hemodynamic compromise requiring cardiopulmonary resuscitation at time of screening
* Suspicion of bowel necrosis (as determined by the implanting physician based on imaging observations, peritoneal signs, surgical exploration, elevated serum lactate levels, low pH, and/or acidosis)
* Clinical or radiographic signs of bowel infarction or gastrointestinal hemorrhage
* Base deficit > -10 mmol/L or -10 mEq/L
* American Society of Anesthesiologists risk class V (i.e., moribund patient not expected to live 24 hours with or without operation) or class VI (a declared brain dead patient whose organs are being removed for donor purposes)
* Previous placement of a thoracic endovascular graft
* Interventional and/or open surgical procedures 30 days prior to the dissection repair
* Planned major interventional and/or open surgical procedures 30 days post the dissection repair
* Systemic infection
* Uncontrollable anaphylaxis to iodinated contrast (patients with allergy to iodinated contrast but not anaphylaxis may be eligible with appropriate pre-medication, as deemed suitable by the Investigator)
* Known allergy(ies) to nitinol and/or polytetrafluoroethylene
* Inability to obtain CT angiograms for follow-up
* Previously diagnosed with Marfan syndrome, Ehlers-Danlos syndrome, or Loeys-Dietz syndrome based on laboratory genetic testing
* Diagnosed with acute myocardial infarction in the 30 days prior to the dissection diagnosis
* Diagnosed with severe and catastrophic neurological complications in the 30 days prior to the dissection diagnosis (namely, obtundation or coma)
* Current Stage 5 end stage chronic kidney disease (eGFR ≤ 15 mL/min)
* History of bleeding disorder (i.e. hemophilia)
* A primary entry tear that extends into the arch or distal to the left subclavian artery
* Need for a total aortic arch replacement and/or repair, or reconstruction, of any part of the arch, and branch vessels (including extra-anatomic bypass of the branch vessels), for any reason as deemed necessary by the Investigator
* Any pathology of mycotic origin
* Aortic fistulous communication with non-vascular structure (e.g., esophagus, bronchial)
* Extensive thrombus or calcifications in the aortic arch, as defined by CTA
* Excessive tortuosity precluding safe passage of the AMDS, as defined by CTA
* Descending thoracic aneurysm involving the proximal third (one-third) of the descending aorta and measuring >45 mm in diameter
* Aortic arch aneurysm >50 mm in diameter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2029-12-06 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint to Assess Incidence of Major Adverse Events | Through 30 days
  Patients experiencing at least one of the following MAEs:
  1. All-cause mortality (ACM)
  2. New disabling stroke
  3. New onset renal failure requiring dialysis
  4. Myocardial infarction (MI)
Primary Endpoint to Assess Distal Anastomotic New Entry (DANE) tears | Through 30 days
  Patients experiencing Distal Anastomotic New Entry (DANE) tears

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Szeto, MD, Principal Investigator — University of Pennsylvania
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory University Medical Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York
  - Northwell, New York, New York
  - Montefiore Einstein Medical, The Bronx, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Ascension Seton/University of Texas, Austin, Texas
  - Baylor College of Medicine/ St. Luke's Medical Center, Houston, Texas
  - Baylor Scott & White The Heart Hospital Plano, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szeto WY, Fukuhara S, Fleischman F, Sultan I, Brinkman W, Arnaoutakis G, Takayama H, Eudailey K, Brinster D, Jassar A, DeRose J, Brown C, Farrington W, Moon MC. A novel hybrid prosthesis for open repair of acute DeBakey type I dissection with malperfusion: Early results from the PERSEVERE trial. J Thorac Cardiovasc Surg. 2025 Jul;170(1):114-123.e3. doi: 10.1016/j.jtcvs.2024.07.059. Epub 2024 Aug 6. PMID 39116932
- [Derived] Brinkman W, Squiers JJ, Jassar A, Fukuhara S, Fleischman F, Takayama H, Sultan I, Arnaoutakis G, Moon MC, Szeto WY; PERSEVERE Investigators. Cerebral malperfusion resolution after repair of acute DeBakey type I dissection with a novel hybrid prosthesis: early results of the PERSEVERE Studydagger. Eur J Cardiothorac Surg. 2025 Jul 1;67(7):ezaf199. doi: 10.1093/ejcts/ezaf199. PMID 40586922